CLINICAL TRIAL: NCT02646995
Title: Lipid Formulation to Increase the Bioavailability of Fatty Acids in Cystic Fibrosis (CF) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 14.18.CLI
Record Dates: First submitted 2015-12-22; First posted 2016-01-06 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): modified lipid formulation
  Interventions: Dietary Supplement: modified lipid formulation
- Control (Active Comparator): fish oil
  Interventions: Dietary Supplement: Fish oil

INTERVENTIONS:
Dietary Supplement: modified lipid formulation — Tested oils will be used in liquid form and encapsulated in soft gelatin capsules.
  Arms: Active
Dietary Supplement: Fish oil — Fish oil will be used in liquid form and encapsulated in soft gelatin capsules.
  Arms: Control

SUMMARY:
The purpose of this trial is to evaluate if the use of a newly developed lipid formulation versus fish oil would better enable the absorption of essential fatty acids after 12 weeks of supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed CF according to established criteria (diagnosis of CF will be based on either two positive sweat chloride tests of >60 mEq/L or the identification of two detectable mutations associated with CF)
2. Exocrine pancreatic insufficiency defined by pathological fecal elastase (<15µg/g) found in the Medical History of the patient
3. Informed consent letter signed and dated by their parents or legal guardians before inclusion in the study, and assent signed and dated by the child if he or she is ≥ 14 years old

Exclusion Criteria:

1. Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for CF or for CF-related conditions within 4 weeks prior to baseline
2. Exposure to another investigational drug or dietary supplements and enteral nutrition containing EPA and docosahexaenoic acid (DHA), Fish or the use of any other supplement containing fish oil within 4 weeks prior to baseline.
3. Treatment with intravenous antibiotics within 4 weeks prior to baseline
4. Newly started oral antibiotic treatment within 4 weeks prior to Baseline
5. History of solid organ or hematological transplantation
6. Ongoing immunosuppressive therapy (other than corticosteroids) within 3 weeks prior to baseline
7. Major complications of lung disease (including massive hemoptysis, pneumothorax, or pleural effusion) within 8 weeks prior to baseline
8. Evidence of pulmonary exacerbation or acute upper or lower respiratory tract infection (including viral illnesses) within 3 weeks prior to baseline
9. Having donated blood or had a transfusion of blood/blood products during the trial and 3 months prior to screening or expected to do so during the study
10. Any bleeding disorders at screening
11. Patient who cannot be expected to comply with the study procedures.
12. Currently participating or having participated in another clinical trial within 8 weeks prior to baseline.
13. Any known food allergy
14. Incapacity to swallow capsules

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Difference of accretion in erythrocytes of eicosapentanoic acid (EPA) between the 2 groups from Baseline to V3 (12 weeks of treatment), as determined by gas chromatography | From Baseline till 12 weeks of treatment (V3)
  determine the accretion in erythrocytes of EPA derived from the modified lipd formulation as compared to EPA from fish oil between the 2 groups after 12 weeks of supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland